CLINICAL TRIAL: NCT02716922
Title: Cervical Cerclage for Singleton Gestations With Short Cervix and Without Prior Preterm Birth
Brief Title: Cerclage for Singletons With Short Cervix Without Prior Preterm Birth
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Gabriele Saccone, Medical Doctor, Federico II University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 33/2016
Record Dates: First submitted 2016-03-06; First posted 2016-03-23 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2016-03

CONDITIONS: Preterm Birth
MeSH Terms: conditions — Premature Birth | interventions — Cerclage, Cervical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cervical cerclage (Experimental): Women randomized to receive cerclage should receive cervical cerclage Cerclage is a circumferential stitch of non-absorbable suture placed around the cervix
  Interventions: Procedure: Cervical cerclage
- No intervention (No Intervention): No cerclage Women randomized to not receive cerclage represent the control arm

INTERVENTIONS:
Procedure: Cervical cerclage — Cerclage is a circumferential stitch of non-absorbable suture placed around the cervix Cerclage type: McDonald Cerclage Suture: Permanent monofilament Pericerclage antibiotics: none Pericerclage tocolytics: none Bed rest: not recommended (in both groups)
  Arms: Cervical cerclage

SUMMARY:
Preterm birth remains the most common cause of perinatal morbidity and mortality. A short cervi- cal length on transvaginal ultrasonography has been shown to be one of the best predictors of preterm birth. In 2005 a meta-analysis by Berghella et al. showed that cervical cerclage does not prevent preterm birth (PTB) in women with short cervical lenght without prior PTB. However maybe the meta-analysis did not reach the statistical significance due to the small sample size

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy (limits the participants to female gender)
* Short cervical length (less than or equal to 25 mm) on second trimester ultrasound at 18-23 6/7 weeks gestation
* 18-50 years of age

Exclusion Criteria:

* Multiple gestation
* Prior spontaneous preterm birth 16-36 6/7 weeks
* Ruptured membranes
* Lethal fetal structural anomaly
* Fetal chromosomal abnormality
* Pessary in place (or planned placement)
* Vaginal bleeding
* Suspicion of chorioamnionitis
* Ballooning of membranes outside the cervix into the vagina or CL = 0 mm on transvaginal ultrasound
* Painful regular uterine contractions
* Placenta previa

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2016-03; Primary Completion 2018-04 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Spontaneous preterm birth rates <34weeks | Less than 34 weeks gestation

SECONDARY OUTCOMES:
Spontaneous preterm birth rates <37, <28 and <24 weeks | Less than 24, 28, and 37 weeks gestation
Type of delivery | Time of delivery
  Cesarean delivery, Spontaneous vaginal delivery, operative vaginal delivery
Spontaneous rupture of membranes | Less than 34 weeks gestation
  Ruptured membranes <34 weeks
Neonatal death | Between birth and 28 days of age
birth weight | Time of delivery
Chorioamnionitis | Time of delivery
  histologic diagnosis of chorioamnionitis
necrotizing enterocolitis | Between birth and 28 days of age
intraventricular hemorrhage | Between birth and 28 days of age
  intraventricular hemorrhage (grade 3 or higher)
respiratory distress syndrome | Between birth and 28 days of age
bronchopulmonary dysplasia | Between birth and 28 days of age
blood-culture proven sepsis | Between birth and 28 days of age
neonatal mortality | Between birth and 28 days of age
  death of a live-born baby within the first 28 days of life
perinatal death | Until 28 days of age
  either fetal mortality or neonatal mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Gabriele Saccone, Napoli, Italy

IPD SHARING:
Plan to Share IPD: No